CLINICAL TRIAL: NCT00702078
Title: Randomised Clinical Study on the Effect of Home-based Treatment of Patients With COPD. Improved Cooperation Between Hospital and Primary Healthcare System.
Brief Title: Home-based Treatment of Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD-HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Community Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17417
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: COPD
Keywords: COPD; home-based treatment; early intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (Other): follow-up according to todays best practice.
  Interventions: Behavioral: usual care
- cooperation (Experimental): Follow-up from the hospital and the primary healthcare in cooperation
  Interventions: Behavioral: closer collaboration between hospital and primary healthcare system

INTERVENTIONS:
Behavioral: closer collaboration between hospital and primary healthcare system — Follow-up from the hospital and the primary healthcare in cooperation
  Arms: cooperation
Behavioral: usual care — follow-up according to todays best practice
  Arms: usual care

SUMMARY:
We want to improve the treatment of patients suffering from COPD (3-4) by early medical intervention in the patients home. A close cooperation between the hospital and the primary healthcare system will hopefully reduce hospitalisation, drug consumption and improve quality of life. Following up from the hospital and the primary healthcare in cooperation may lead to earlier detection and treatment of exacerbations in COPD.

The main outcome variable will be number of hospitalizations assessed simply by counting. The second objective will be Quality of life and activation assessed by different questionnaires included in St.George´s Respiratory Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD (III-IV)
* receive help from homecare nurse
* not suffering from any other serious disease, with expected lifespan less than 6 months

Exclusion Criteria:

-

Max Age: 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations | 2011

SECONDARY OUTCOMES:
quality of life | 2011
lung function | 2011
use of medication | 2011
cost-effectiveness | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hildur Henriksen, MD,PhD, Study Chair — St.Olavs Hospital HF
Locations (1):
- Dept. of Lung Diseases, St.Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Titova E, Salvesen O, Bentsen SB, Sunde S, Steinshamn S, Henriksen AH. Does an Integrated Care Intervention for COPD Patients Have Long-Term Effects on Quality of Life and Patient Activation? A Prospective, Open, Controlled Single-Center Intervention Study. PLoS One. 2017 Jan 6;12(1):e0167887. doi: 10.1371/journal.pone.0167887. eCollection 2017. PMID 28060921